CLINICAL TRIAL: NCT01826617
Title: Configuration of a New Prostate Disease Nomogram Predicting Prostate Biopsy Outcome Correlating Clinical Indicators Among Asian Adult Males With Elevated Prostate Specific Antigen (PSA)
Brief Title: Configuration of a New Prostate Disease Nomogram Predicting Prostate Biopsy Outcome
Status: Completed | Type: Observational
Sponsor: St. Luke's Medical Center, Philippines (Other)
Responsible Party: Principal Investigator, Michael E. Chua, Medical Staff Urologist, St. Luke's Medical Center, Philippines
Other Study IDs: CT-13008; SLMC CT-13008 (Other: SLMC CT-13008)
Record Dates: First submitted 2013-04-01; First posted 2013-04-08 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Prostate Cancer; Prostatitis; Benign Prostatic Hyperplasia
Keywords: Prostate Disease Nomogram; Asian Men
MeSH Terms: conditions — Prostatic Neoplasms; Prostatitis; Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- Prostate Cancer- Indolent type: Patients diagnosed with Indolent type will be classified according to Epstein Criteria on histopathology results and National Comprehensive Cancer Network (NCCN) guideline recommended classification
- Prostate cancer- aggressive type: Patients diagnosed with aggressive type will be classified according to Epstein criteria on final histopathology findings and NCCN guideline recommended classification
- Acute Prostatitis: Patient diagnosed with Acute prostatitis- according to histopathology description of Biopsy result
- Chronic Prostatitis: Patient diagnosed with Chronic prostatitis- according to histopathology description of Biopsy result
- Benign Prostatic Nodular Hyperplasia: Patient diagnosed with Benign Prostatic Nodular Hyperplasia- according to histopathology description of Biopsy result

SUMMARY:
This study will identify significant clinical parameters and individual risk factors related to certain prostate disease (BPH, prostatitis and prostate cancer). With the identified important correlations, a locally generated bias free nomogram will be constructed for predicting prostate biopsy outcome among Asian men with indications for prostate biopsy. While this study will evaluate the accuracy and predictive value of this novel prostate disease nomogram.

DETAILED DESCRIPTION:
This is a cross-sectional study prospectively collecting data from all patients who had their first Transrectal ultrasound (TRUS) prostate biopsy at the Stone and Prostate Treatment Center of St. Luke's Medical Center-Quezon City . Data will be collected uniformly for the purpose of building a clinical care prostate biopsy database. The indication for prostate biopsy is either a suspicious DRE findings or elevated Prostate specific antigen (PSA) level (>4.0ng/ml) or both. The clinical information gathered will include the 1. Identified risk factors (age, family history, race, Body Mass Index (BMI) - kg/cm2, prostatitis, and medications) 2. Clinical indicators of prostatic diseases (abnormal digital rectal examination, hypoechoic lesion on transrectal ultrasound), and 3. PSA (ng/ml) and its derivatives (age-specific PSA, PSA density, PSA velocity, Free PSA percentage). (Refer to Data Collection Form). Basic demographic data such as patient's height and weight will be measured using standard weight scale (Detecto 439 Mechanical Scale with Height rod, Webb City MO, USA). A urologist member of the team will perform DIgital Rectal Exam (DRE) on all patients before or after the TRUS. Serum free and total PSA level is measured at the Institute of Pathology using Siemens ADVIA Centaur Free PSA and PSA (Seimens Healthcare Diagnostics, USA) within a month prior to the prostate biopsy. Prior to prostate biopsy, the prostate will be scanned using a biplanar 7.5 Megahertz probe (GE Medical Systems Kretz Ultrasound, Zipf, Austria. Prostate volume is measured by a radiology technician [member of the staff team] of the center using the transverse and sagittal planes with the standard equation of measurement for prolate ellipsoid [width (w) x height (h) x length (l) x 0.523].

All prostate biopsy will uniformly required 12 cores (extended scheme) or more prostate tissue strips under ultrasound guidance with Fr 18 25cm biopsy device (Bard Urological, US), it is performed systematically to covers lateral and medial aspects of the apex, midgland and base of the right and left prostate lobes. Two additional biopsies are obtained if the ultrasound image or DRE findings indicate suspect areas.

All acquired specimens are placed in a formalin-filled container and sent for histopathologic examination. All specimens are examined by at least 2 board-certified pathologists at the Institute of Pathology to determine the presence of inflammation (acute/chronic prostatitis), other disease entity, or carcinoma (if positive for carcinoma, reading include grade using Gleason score, cancer length in biopsy specimen, percent of cancer involvement. All pathologists are blinded from the clinical indicators of the patients. An intermediate result is further subjected to immunohistostaining for a definitive conclusion. At least two pathologists are required to release the final report.

Data collection and extraction will use the pre-tested and standardized form. All collected forms will be submitted to the Clinical Information Service of St. Luke's Medical Center for encoding and preliminary analysis of incidence and prevalence. Additional analysis will be sent to a third party statistician for validation and reliability check.

Confidentiality of all data acquired will be assured. All patient record will be coded in the database as PIN. Patient name will not be included for encoding into the databank. Only the investigator team and clinical information service section of St. Luke's Medical Center will have access to the data set encoded. Hospital policy on safekeeping of the hospital record will be strictly followed and stored by Medical Record section of the medical center.

ELIGIBILITY:
Inclusion Criteria:

* All patients who had their first Transrectal ultrasound (TRUS) prostate biopsy at the Stone and Prostate Treatment Center of St. Luke's Medical Center-Quezon City . The indication for prostate biopsy is either a suspicious DRE findings or elevated PSA level (>4.0ng/ml) or both.

Exclusion Criteria:

* non-Asian patient
* incomplete data provided and patients refused to provide required data
* Prostate specific antigen done other than St. Luke's Medical Center
* did not consent for biopsy procedure

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a cross-sectional study prospectively collecting data from all patients who had their first Transrectal ultrasound (TRUS) prostate biopsy at the Stone and Prostate Treatment Center of St. Luke's Medical Center-Quezon City . Data will be collected uniformly for the purpose of building a clinical care prostate biopsy database. The indication for prostate biopsy is either a suspicious DRE findings or elevated PSA level (>4.0ng/ml) or both.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2010-12; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Incidence of prostate cancer (indolent vs aggressive type) | 1 year
  Incidence of new diagnosed prostate cancer among patients with indication presented for first TRUS prostate biopsy at stone and prostate treatment center.
Incidence of prostatitis (acute vs chronic) | 1 year
  Incidence of new diagnosed prostatitis among patients with indication presented for first TRUS prostate biopsy at stone and prostate treatment center.
Incidence of nodular hyperplasia (benign prostatic hyperplasia) | 1 year
  Incidence of new diagnosed nodular hyperplasia (benign prostatic hyperplasia) among patients with indication presented for first TRUS prostate biopsy at stone and prostate treatment center.

SECONDARY OUTCOMES:
Incidence of patient with synchronous occurrence of prostate diseases (benign prostatic hyperplasia, prostatitis, prostate cancer) | 1 year
  Incidence of new diagnosed synchronous occurrences of prostate diseases (benign prostatic hyperplasia, prostatitis, prostate cancer) among patients with indication presented for first TRUS prostate biopsy at stone and prostate treatment center.

OTHER OUTCOMES:
Mean Age of patients with prostate cancer (PCA) or Prostatitis or BPH | 1 year
Mean PSA value of patients with PCA, or Prostatitis or BPH | 1 year
Mean BMI of patients with PCA, or Prostatitis or BPH | 1 year
Mean PSA density of patients with PCA, or Prostatitis or BPH | 1 year
Mean PSA velocity of patients with PCA, or Prostatitis or BPH | 1 year
Mean percent free PSA of patients with PCA, or Prostatitis or BPH | 1 year
Prevalence of positive family History of patients with Prostate cancer, or Prostatitis or BPH | 1 year
Prevalence of abnormal DRE of patients with PCA, or Prostatitis or BPH | 1 year
Prevalence of TRUS findings of patients with PCA, or Prostatitis or BPH | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Michael E. Chua, MD, Principal Investigator — St. Luke's Medical Center, Philippines
Locations (1):
- Stone and Prostate Treatment Center- St. Luke's Medical Center, Philippines, Quezon City, National Capital Region, Philippines